CLINICAL TRIAL: NCT06820463
Title: A Phase 2, Open-Label, Randomized, Master Protocol Study to Evaluate Safety and Efficacy of Multiple Treatment Combinations With Telisotuzumab Adizutecan in Subjects With Metastatic Colorectal Cancer
Brief Title: A Study to Evaluate the Adverse Events, and Efficacy of Intravenous (IV) of Telisotuzumab Adizutecan in Combination With IV Oxaliplatin, Fluorouracil, Folinic Acid/Leucovorin, Bevacizumab, Panitumumab in Adult Participants With Metastatic Colorectal Cancer
Acronym: AndroMETa-CRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24-533; EU CT (Other: 2024-512981-33-00)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; AndroMETa-CRC-533; Telisotuzumab Adizutecan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Oxaliplatin; Leucovorin; Bevacizumab; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Substudy 1: Dose Escalation Telisotuzumab Adizutecan (Experimental): Participants will receive various doses of telisotuzumab adizutecan in combination with a fixed dose of fluorouracil, leucovorin, and oxaliplatin (FOLFOX) and bevacizumab as part of the approximately 6 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Bevacizumab
- Substudy 1: Dose Expansion Telisotuzumab Adizutecan High Dose (Experimental): Participants will receive the high dose of telisotuzumab adizutecan determined in the dose expansion arm in combination with a fixed dose of FOLFOX and bevacizumab as part of the approximately 6 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Bevacizumab
- Substudy 1: Dose Expansion Telisotuzumab Adizutecan Low Dose (Experimental): Participants will receive the low dose of telisotuzumab adizutecandetermined in the dose expansion arm in combination with a fixed dose of FOLFOX and bevacizumab as part of the approximately 6 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Bevacizumab
- Substudy 1: Dose Expansion Compatator (Experimental): Participants will receive a fixed dose of FOLFOX and bevacizumab as part of the approximately 6 year study duration.
  Interventions: Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Bevacizumab
- Substudy 2: Dose Escalation Telisotuzumab Adizutecan (Experimental): Participants will receive various doses of telisotuzumab adizutecan in combination with a fixed dose of fluorouracil (5-FU) and leucovorin (LV) and panitumumab as part of the approximately 6 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Fluorouracil; Drug: Leucovorin; Drug: Panitumumab
- Substudy 2: Dose Expansion Telisotuzumab Adizutecan High Dose (Experimental): Participants will receive the high dose of telisotuzumab adizutecan determined in the dose expansion arm in combination with a fixed dose of 5-FU/LV and panitumumab as part of the approximately 6 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Fluorouracil; Drug: Leucovorin; Drug: Panitumumab
- Substudy 2: Dose Expansion Telisotuzumab Adizutecan Low Dose (Experimental): Participants will receive the low dose of telisotuzumab adizutecan determined in the dose expansion arm in combination with a fixed dose of 5-FU/LV and panitumumab as part of the approximately 6 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Fluorouracil; Drug: Leucovorin; Drug: Panitumumab
- Substudy 2: Dose Expansion Compatator (Experimental): Participants will receive a fixed dose of FOLFOX and panitumumab as part of the approximately 6 year study duration.
  Interventions: Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Panitumumab

INTERVENTIONS:
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion
  Arms: Substudy 1: Dose Escalation Telisotuzumab Adizutecan; Substudy 1: Dose Expansion Telisotuzumab Adizutecan High Dose; Substudy 1: Dose Expansion Telisotuzumab Adizutecan Low Dose; Substudy 2: Dose Escalation Telisotuzumab Adizutecan; Substudy 2: Dose Expansion Telisotuzumab Adizutecan High Dose; Substudy 2: Dose Expansion Telisotuzumab Adizutecan Low Dose
Drug: Fluorouracil — IV Infusion; IV Injection
Drug: Oxaliplatin — IV Infusion
  Arms: Substudy 1: Dose Escalation Telisotuzumab Adizutecan; Substudy 1: Dose Expansion Compatator; Substudy 1: Dose Expansion Telisotuzumab Adizutecan High Dose; Substudy 1: Dose Expansion Telisotuzumab Adizutecan Low Dose; Substudy 2: Dose Expansion Compatator
Drug: Leucovorin — IV Infusion; IV Injection
Drug: Bevacizumab — IV Infusion
  Arms: Substudy 1: Dose Escalation Telisotuzumab Adizutecan; Substudy 1: Dose Expansion Compatator; Substudy 1: Dose Expansion Telisotuzumab Adizutecan High Dose; Substudy 1: Dose Expansion Telisotuzumab Adizutecan Low Dose
Drug: Panitumumab — IV Infusion
  Arms: Substudy 2: Dose Escalation Telisotuzumab Adizutecan; Substudy 2: Dose Expansion Compatator; Substudy 2: Dose Expansion Telisotuzumab Adizutecan High Dose; Substudy 2: Dose Expansion Telisotuzumab Adizutecan Low Dose

SUMMARY:
CRC is the third most common type of cancer diagnosed worldwide with developed countries at highest risk. The purpose of this study is to assess adverse events and change in disease activity when telisotuzumab adizutecan is given in combination with oxaliplatin, fluorouracil (5FU), leucovorin (LV) (FOLFOX), and bevacizumab or panitumumab.

Telisotuzumab adizutecan is an investigational drug being developed for the treatment of mCRC. Fluorouracil and leucovorin are drugs approved for the treatment of mCRC. This study will be divided into two stages, with the first stage treating participants with increasing doses of telisotuzumab adizutecan with FOLFOX and bevacizumab or 5FU/LV and panitumumab until the dose reached is tolerable and expected to be efficacious. Participants will then be randomized into 3 groups called treatment arms where one group will receive one of two optimized doses of telisotuzumab adizutecan from the dose escalation phase with FOLFOX and bevacizumab or 5FU/LV and panitumumab, or a comparator of FOLFOX and bevacizumab or panitumumab. Approximately 390 adult participants with mCRC will be enrolled in the study in 100 sites worldwide.

In the dose escalation stage participants will be treated with increasing intravenous (IV) doses of telisotuzumab adizutecan with FOLFOX and bevacizumab or 5FU/LV and panitumumab until the dose reached is tolerable and expected to be efficacious. In the dose optimization stage participants will be receive FOLFOX or receive 5FU/LV, but with one of two optimized doses of telisotuzumab adizutecan, or a comparator of FOLFOX and bevacizumab/pantitumumab. The study will run for a duration of approximately 6 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Laboratory values meeting the criteria within the protocol.
* Has measurable disease per response evaluation criteria in solid tumors (RECIST) v1.1.

Exclusion Criteria:

* Prior systemic regimen containing c-Met targeting agent(s) (e.g., antibody, antibody drug conjugate, bispecific) and/or any topoisomerase inhibitor(s) (e.g., irinotecan).
* History of other malignancies within 5 years prior to screening, except for malignancies with a negligible risk of metastasis or death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) as Assessed by the Investigator confirmed complete response (CR) or partial response (PR) as assessed by the investigator per response evaluation criteria in solid tumors (RECIST), version 1.1. | Up to 24 Weeks
  OR is defined as confirmed CR or PR as assessed by the investigator per RECIST, version 1.1.
Number of Participants with Adverse Events (AE)s | Up to Approximately 6 Years
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by the Investigator | Up to 22 Months
  PFS is defined as the time from the first dose of study treatment to the first occurrence of radiographic progression based on RECIST version 1.1 as determined by the investigator or death from any cause, whichever occurs earlier.
Duration of Response (DOR) as Assessed by the investigator | Up to 14 Months
  DOR is defined as the time from the first documented CR or PR to the first occurrence of radiographic progression per RECIST v1.1 as determined by the investigator or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to Approximately 6 Years
  OS is defined as the time from first dose of study treatment to the event of death from any cause.
Disease Control (DC) as Assessed by the Investigator | Up to Approximately 6 Years
  DC is defined as best overall response of confirmed CR or confirmed PR, or stable disease (SD) based on RECIST, version 1.1 as determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (41):
- United States (10):
  - City of Hope National Medical Center /ID# 270255, Duarte, California
  - Yale New Haven Hospital /ID# 270565, New Haven, Connecticut
  - Hope And Healing Cancer Services /ID# 271562, Hinsdale, Illinois
  - Dana-Farber Cancer Institute /ID# 270624, Boston, Massachusetts
  - Saint Lukes Hospital of Kansas City /ID# 270633, Kansas City, Missouri
  - Nebraska Cancer Specialists - Omaha - Wright Street /ID# 271646, Omaha, Nebraska
  - University of North Carolina Medical Center /ID# 267786, Chapel Hill, North Carolina
  - Oncology Hematology Care - Eastgate /ID# 271493, Cincinnati, Ohio
  - Texas Oncology - Austin Midtown /ID# 271354, Austin, Texas
  - Texas Oncology - Deke Slayton Cancer Center /ID# 271355, Webster, Texas
- Australia (5):
  - Macquarie University /ID# 271514, Sydney, New South Wales
  - Mater Hospital Brisbane /ID# 270694, South Brisbane, Queensland
  - The Queen Elizabeth Hospital /ID# 270693, Woodville, South Australia
  - Austin Health /ID# 270692, Heidelberg, Victoria
  - One Clinical Research /ID# 270695, Nedlands, Western Australia
- Medizinische Universitaet Wien /ID# 268872, Vienna, Austria
- Czechia (2):
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 268773, Hradec Králové, Hradec Kralove
  - Thomayerova nemocnice /ID# 269632, Prague, Praha, Hlavni Mesto
- France (3):
  - Chu De Lille - Hopital Claude Huriez /ID# 270222, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Poitiers /ID# 270225, Poitiers, Nouvelle-Aquitaine
  - Hôpital Européen Georges Pompidou /ID# 270224, Paris
- Greece (2):
  - St. Luke's Hospital S.A. /ID# 269963, Panórama, Thessaloniki
  - Theagenio Cancer Hospital /ID# 269640, Thessaloniki
- Israel (5):
  - Tel Aviv Sourasky Medical Center /ID# 268010, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 268006, Haifa
  - Shaare Zedek Medical Center /ID# 268009, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 268007, Jerusalem
  - Rabin Medical Center /ID# 268008, Petah Tikva
- Japan (4):
  - National Cancer Center Hospital East /ID# 270114, Kashiwa-shi, Chiba
  - St Marianna University School Of Medicine /ID# 270111, Kawasaki-shi, Kanagawa
  - Tohoku University Hospital /ID# 270966, Sendai, Miyagi
  - National Cancer Center Hospital /ID# 270112, Chuo-Ku, Tokyo
- Pan American Center for Oncology Trials /ID# 268809, Rio Piedras, Puerto Rico
- Spain (2):
  - Hospital Universitario Marques de Valdecilla /ID# 269732, Santander, Cantabria
  - Hospital Universitario Vall de Hebron /ID# 270191, Barcelona
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 269726, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 269717, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 269724, Kaohsiung City
  - National Cheng Kung University Hospital /ID# 270835, Tainan
  - Taipei Veterans General Hospital /ID# 269718, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 269725, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-533